CLINICAL TRIAL: NCT06588764
Title: Modified Deep Lateral Wall Decompression and/or Deep Medial Wall Decompression for Moderate-to-severe Grave's Ophthalmopathy: a Prospective Study
Brief Title: Modified Orbital Decompression in the Treatment of Moderate-to-severe Grave's Ophthalmopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huasheng Yang, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: yanghs20240821
Record Dates: First submitted 2024-08-27; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Graves Ophthalmopathy; Surgery
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Modified deep lateral and/or medial wall decompression in Moderate-to-severe Graves' Orbitopathy
  Interventions: Procedure: modified deep lateral and/or medial wall decompression

INTERVENTIONS:
Procedure: modified deep lateral and/or medial wall decompression — Modified deep lateral orbital wall decompression is based on traditional outer wall decompression with combined abrasion of the deep outer orbital wall (including the greater pterygoid wing) to achieve adequate enlargement of the orbital cavity.

SUMMARY:
To investigate the efficacy and safety of modified deep lateral wall decompression and/or medial wall decompression for Moderate-to-severe Grave's Ophthalmopathy.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the effectiveness and complications of modified deep lateral wall decompression and medial wall decompression, in order to develop a standardized technical approach to the treatment of Moderate-to-severe Grave's Ophthalmopathy.

ELIGIBILITY:
Inclusion Criteria:

1. EUGOGO/NOSPECS grade was moderate-to-severe thyroid associate ophthalmopathy;
2. CAS≤3 score;
3. stable thyroid function for at least 6 months;
4. able and willing to participate in clinical trials and ensure regular follow-up;

Exclusion Criteria:

1. any uncontrollable clinical problems (severe mental, neurological, cardiovascular, respiratory and other systemic diseases and malignant tumors);
2. B-ultrasound or CT, MRI found other diseases causing exophthalmos (intraorbital space occupying lesion, inflammatory pseudotumor, neurofibroma, etc.);
3. uveitis, glaucoma, high myopia, diabetic retinopathy and other eye diseases
4. those who were considered by the researchers to be excluded

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
best corrected visual acuity (BCVA) | within 24 weeks of surgery
  Using Snellen scale, decimal fraction

SECONDARY OUTCOMES:
value of Hertel | within 24 weeks of surgery
  as measured using a Hertel exophthalmometer, to describe the degree of exophthalmos
the mean deviation value of visual field (VF) | 24 weeks after surgery
  The mean deviation (MD) gives an overall value of the total amount of visual field loss, with normal values typically within 0dB to -2dB. The mean deviation value of visual field (VF) was examined by HFA (Humphrey II, Carl-Zeiss, Dublin, CA).
pattern standard deviation value of visual field | within 24 weeks of surgery
  The pattern standard deviation (PSD) can filter out the decrease in visual acuity caused by turbidity of the dioptric interstitial. The pattern standard deviation (PSD) was examined by HFA (Humphrey II, Carl-Zeiss, Dublin, CA).
the P100 latency of pattern visual evoked potential (PVEP) | within 24 weeks of surgery
  The visual stimulus was a pattern reversal checkerboard displayed on a black and white monitor placed 105 cm from the patient. The wave latency of P100 was recorded.
N75-p100 amplitude of PVEP | within 24 weeks of surgery
  Wave amplitude difference between N75-P100 peak and trough.
clinical activity score (CAS) | within 24 weeks of surgery
  The CAS is a 7-item description of clinical activity, including: 1. Spontaneous orbital pain; 2. Gaze evoked orbital pain; 3. Eyelid swelling that is considered to be due to active (inflammatory phase) thyroid eye disease/ Graves' Ophthalmopathy or Orbitopathy (TED/GO); 4. Eyelid erythema; 5. Conjunctival redness that is considered to be due to active (inflammatory phase) TED/GO (ignore "equivocal" redness); 6. Chemosis; 7. Inflammation of caruncle or plica.
volume of adipose tissue | during the surgery
  Prolapsing extraconal and intraconal orbital fat were resected from the orbital margin deep into the intraconal apex. The desired volume of adipose tissue was measured intraoperatively using 5 or 10 cc syringe.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No